CLINICAL TRIAL: NCT03315390
Title: PTSD After ICU Survival - Caring for Patients With Traumatic Stress Sequelae Following Intensive Medical Care - a Multi-Center, Observer-blinded, Randomized, Controlled Trial With a Psychological Intervention
Brief Title: PTSD After ICU Survival - Caring for Patients With Traumatic Stress Sequelae Following Intensive Medical Care
Acronym: PICTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: German Research Foundation (Other); University of Konstanz (Other)
Responsible Party: Principal Investigator, Jochen Gensichen, Direktor am Institut für Allgemeinmedizin, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GE 2073/8-1
Record Dates: First submitted 2017-10-10; First posted 2017-10-20 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: post-traumatic stress, primary health care, stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic

STUDY DESIGN:
Intervention Model Description: multi-center, observer-blinded, randomized, controlled trial with complex psychological intervention
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-group (Experimental): Narrative Exposure Therapy (NET): for GP-practice adapted version of narrative exposure therapy during 3 sessions (à 45 minutes)
  Interventions: Other: "Narrative Exposure Therapy"-oriented intervention
- iTAU group (Active Comparator): Improved Treatment-as-usual: 3 GP consultations with patients according to guidelines and adapted to patients' needs
  Interventions: Other: improved treatment as usual (iTAU)

INTERVENTIONS:
Other: "Narrative Exposure Therapy"-oriented intervention — Narrative Exposure Therapy (NET) in an Primary-care adapted Version in 3 sessions (S) 6 weeks (S1), 8 weeks (S2) and 12 weeks (S3) after baseline data collection at T0.
  Arms: Intervention-group
Other: improved treatment as usual (iTAU) — improved standard primary care for PTSD according to Guidelines, customized to patients' needs and symptoms during 3 consultations between T0 and T1
  Arms: iTAU group

SUMMARY:
During the PICTURE trial a short narrative therapy (narrative exposure therapy adapted for primary care) for patients with posttraumatic stress disorder (PTSD) after intensive care treatment is to be carried out by their general practitioner (GP). During regular practice hours, this is often difficult. For this reason, we are investigating whether the regular treatment can be improved by a specially trained GP.

The aim of the study is to investigate the effects and applicability of a short version of an established narrative therapy for patients with posttraumatic stress disorders after intensive medical treatment.

Three months after discharge from the intensive care unit, the diagnosis of a PTSD symptoms is verified and the patients are randomized into two groups.

In the treatment group, the physician will perform three 45-minute therapy sessions with the patient within 6 weeks. During the first session a list of the most intense events - both positive and negative - in the life of the patient is drawn on the basis of a life line, with the stay at the intensive care unit being one of these events. The second session deals with the experience during intensive care in detail, led by the GP. During the third session, another event from the patient's life will be discussed in the same manner. This way, the different components (cognitions, emotions, body reactions, context information) can be reconnected and classified into the patient's own biography. Between the therapy sessions, a conversation between the GP and the psychologist will take place to support the GP during the therapy. In order to monitor the patient's safety and compliance, standardized telephone calls between the patient and the GP practice are regularly carried out every 2-3 weeks in between therapy sessions up to the first data collection after 6 months (T1).

In the control group there are three doctor-patient contacts, too, which content is based on the patient's symptoms. This group thus receives the standard therapy which is customary in practice.

DETAILED DESCRIPTION:
The treatment of patients with posttraumatic stress disorder (PTSD) in general practice is usually symptom-oriented and does not necessarily involve a proactive approach. Instead, PTSD is often not verbalized, and patients are treated symptomatically or referred to specialists / psychologists, often associated with long waiting times.

We are conducting this trial to investigate a short, narrative exposure therapy (NET) adapted for the use by general practitioners (GPs) in patients with PTSD symptoms after intensive care treatment. NET is the only method that has proved to be successful in PTSD patients, even when used by paramedics, nurses or local counselors, and is therefore also suitable for physicians without extensive psychological training The aim of our study is 1) to examine the feasibility and safety of a NET-oriented therapy in primary care, and 2) to examine the effects of the NET-oriented therapy in comparison to standard care by collecting results 6 and 12 months after diagnosis.

The intervention is being investigated in a randomized controlled, observer-blinded multicenter study with two arms. 318 patients (and their GPs) are included in 2 locations (Munich & Berlin) in Germany.

3 months after discharge from intensive care unit, the diagnosis of PTSD symptoms in participants is verified by the GP and patients are randomly assigned to either treatment group or the control group.

In the treatment group, the GPs receive training in executing narrative exposure therapy by specialized psychologists. The doctors of this group will hold three 45-minute therapy sessions with their patient within 6 weeks. During the first session a list of the most intense events - both positive and negative - is drawn up in the life of the patient on the basis of a life line, with the stay at the intensive care unit being one of these events. During the second session the experience in the intensive care unit will be discussed in detail, led by the GP. During the third session, another event from the patient's life is dealt with in the same manner. This way, the different components (cognitions, emotions, body reactions, context information) can be reconnected and classified into the patient's own biography. Between therapy sessions, the GP and the psychologist will schedule a conversation for support and supervision of the GP during the therapy. In order to monitor the patient's safety and compliance, standardized telephone calls between the patient and the GP's practice are regularly carried out every two-three weeks in between the therapies sessions and up to the first data collection after six months (T1).

In the control group, the GPs receive training in treatment of PTSD according to guidelines. In this group, there are also 3 consultations between GP and patient. However, the content of these consultations is based on the patient's symptoms. This group thus receives the standard therapy which is customary in practice.

The data necessary for the evaluation of the intervention is collected 6 and 12 months after the first GP appointment, during which the diagnosis was verified.

ELIGIBILITY:
Patients:

Inclusion Criteria: Symptoms for Posttraumatic Stress disorder (PDS-5 [2016] Score ≥ 15 (20-item Posttraumatic Diagnostic Scale for the Diagnostic and Statistical Manual of Mental Disorders (DSM) -5)); written informed consent of the patient is present; sufficient knowledge of the German language in word and writing; patients must be able to follow study instructions and likely to attend and complete all required visits and telephone surveys.

Exclusion criteria: physical or psychiatric condition which may put the patient at risk, may confound the trial results or may interfere with the patient's participation in this trial; known or persistent abuse of medication, drugs or alcohol as assessed by the GP; major depression (PHQ-9 score ≥ 23), acute suicidality, life expectancy <6 months at T0; already receiving another psychotherapeutic trauma therapy such as Eye Movement Desensitization and Reprocessing (EDMR) or Cognitive behavioral therapy (CBT) at T0; any neuroleptic, anticholinergic or anti-epileptic drugs as permanent medication for specific psychiatric disease within the last two weeks prior to baseline;

GPs:

Inclusion criteria: providing family doctor services for ≥ 2 years within the German statutory health care system, holding a certificate for "Basic Psychosomatic Care" (German Medical Association 2001), alternatively, GP has to be a family doctor within the German statutory health care system for ≥ 5 years with adequate psychological, psychosomatic or psychiatric qualification; informed consent of the GP is present Exclusion criteria: GPs: > 80% of patients with a specific mental condition

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2018-10-21 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Stress | from baseline data collection to 6-month follow-up
  absolute change in posttraumatic stress symptoms as measured by the Posttraumatic Stress Diagnostic Scale (PDS-5) total severity score; each of the 20 items refers to symptoms experienced in the past month and is answered on a 5-point Likert scale ranging from 0 (not at all) to 4 (more than 5 times per week/severe), total score range 0 - 80 points

SECONDARY OUTCOMES:
Posttraumatic Stress | from baseline data collection to 12-month follow-up
  absolute change in posttraumatic stress symptoms as measured by the Posttraumatic Stress Diagnostic Scale (PDS-5) total severity score; each of the 20 items refers to symptoms experienced in the past month and is answered on a 5-point Likert scale ranging from 0 (not at all) to 4 (more than 5 times per week/severe), total sum score range 0 - 80 Points, with a high score indicating severe impairment
Depression | from baseline data collection to 6-month and 12-month follow-up
  absolute change in depressive symptoms experienced over the last 2 weeks as measured by the Patient Health Questionnaire (PHQ)-9 total score; each of the 9 items items is scored from 0 (not at all) to 3 (nearly every day); total sum score range from 0 to 27 points, with a high score indicating severe impairment
Anxiety | from baseline data collection to 6-month and 12-month follow-up
  absolute change in anxiety severity and impairment as measured by the Overall Anxiety Severity and Impairment Scale (OASIS) total score; there are 5 response options for each of the 5 items, which are coded from 0 to 4; total sum score range from 0 (no anxiety) to 20 points, with a high score indicating severe impairment
Patient's self-rated health | from baseline data collection to 6-month and 12-month follow-up
  absolute change in health-related quality of life as measured by the EuroQol - 5 Dimensions (5D) - 5 Level (EQ-5D-5L) Visual Analogue Scale (VAS); the EQ-5D-5L VAS is a thermometer-like rating scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Disability | from baseline data collection to 6-month and 12-month follow-up
  absolute change in disability as measured by the World Health Organization Disability Assessment Schedule (WHODAS) 2.0 - short version total score (12-item Version); range from 0 to 100, with higher scores indicating higher Levels of disability
Patient Activation Measure | from baseline data collection to 6-month and 12-month follow-up
  absolute change in active participation of patients and the self-management of their state of health as measured by the Patient Activation Measure-13 (PAM-13) total score (13-items); each item scores from 1 to 4 (1 = strongly disagree, 2= disagree, 3=agree, 4= strongly agree; for the fifth item only additionally 5= not applicable); Evaluation is made by adding the raw values with a range of 13 - 52; sum-scale will be calibrated to a 0 to 100 metric
Cost-effectiveness | from baseline data collection to 6-month and 12-month follow-up
  absolute change in health-related costs as measured by the modified Client Sociodemographic and Service Receipt Inventory (CSSRI) based on direct and indirect costs

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Gensichen, Prof. Dr., Principal Investigator — Institut für Allgemeinmedizin, LMU München
Locations (2):
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Ludwig-Maximilians-Universität München, München

IPD SHARING:
Plan to Share IPD: Yes
Yes. Deidentified participant data, data dictionary. The data will only be made available to scientific institutions that submit a methodologically meaningful evaluation proposal. Furthermore, applicants must sign a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available 01-01-2025.
Access Criteria: Requests to be sent to the Principal Investigator for access to the anonymous participant data. Data will be made available to researchers whose proposed use of the data has been approved. Data will be made available for the advancement of medical research in line with a Data Use Agreement.

REFERENCES:
- [Derived] Gensichen J, Schmidt KFR, Sanftenberg L, Kosilek RP, Friemel CM, Beutel A, Dohmann J, Heintze C, Prescott HC, Reips UD, Schauer M, Lindemann D, Brettschneider C, Dreischulte T, Zwissler B, Elbert T; PICTURE study group. Effects of a general practitioner-led brief narrative exposure intervention on symptoms of post-traumatic stress disorder after intensive care (PICTURE): multicentre, observer blind, randomised controlled trial. BMJ. 2025 May 7;389:e082092. doi: 10.1136/bmj-2024-082092. PMID 40335079
- [Derived] Beutel A, Sanftenberg L, Friemel CM, Kosilek RP, Schauer M, Elbert T, Reips UD, Schubert T, Gehrke-Beck S, Schmidt K, Gensichen J; PICTURE study group. Patient perspectives on stress after ICU and a short primary care based psychological intervention - results from a qualitative sub-study of the PICTURE trial. BMC Prim Care. 2025 Jan 15;26(1):12. doi: 10.1186/s12875-024-02698-6. PMID 39815198
- [Derived] Gensichen J, Schultz S, Adrion C, Schmidt K, Schauer M, Lindemann D, Unruh N, Kosilek RP, Schneider A, Scherer M, Bergmann A, Heintze C, Joos S, Briegel J, Scherag A, Konig HH, Brettschneider C, Schulze TG, Mansmann U, Linde K, Luhmann D, Voigt K, Gehrke-Beck S, Koch R, Zwissler B, Schneider G, Gerlach H, Kluge S, Koch T, Walther A, Atmann O, Oltrogge J, Sauer M, Schnurr J, Elbert T; PICTURE Study Group. Effect of a combined brief narrative exposure therapy with case management versus treatment as usual in primary care for patients with traumatic stress sequelae following intensive care medicine: study protocol for a multicenter randomized controlled trial (PICTURE). Trials. 2018 Sep 10;19(1):480. doi: 10.1186/s13063-018-2853-7. PMID 30201053

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT03315390/SAP_002.pdf